CLINICAL TRIAL: NCT04172792
Title: Safety and Tolerability of Fat-rich vs. Carbohydrate-rich High-caloric Food Supplements in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Safety and Tolerability Ultra-high-caloric Food Supplements in Amyotrophic Lateral Sclerosis (ALS)
Acronym: TOLCAL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Christian Ludolph, Prof. (Other)
Collaborators: Nutritia GmbH, 91052 Erlangen, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Albert Christian Ludolph, Prof., Prof. Dr., University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOLCAL
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- high-caloric fatty diet (Active Comparator): intake of 405 kcal (45g fat) per day in addition to normal food intake
  Interventions: Dietary Supplement: high-caloric fatty diet
- ultra-high-caloric fatty diet (Experimental): intake of 810 kcal (90g fat) per day in addition to normal food intake
  Interventions: Dietary Supplement: ultra-high-caloric fatty diet
- ultra-high-caloric carbohydrate-rich diet (Experimental): intake of 900 kcal (111.4g carbohydrate, 34.9g fat, 36.0g protein) in addition to normal food intake
  Interventions: Dietary Supplement: ultra-high-caloric carbohydrate-rich diet
- control (No Intervention): normal food intake (no intervention)

INTERVENTIONS:
Dietary Supplement: high-caloric fatty diet — see arm/group description
  Arms: high-caloric fatty diet
Dietary Supplement: ultra-high-caloric fatty diet — see arm/group description
  Arms: ultra-high-caloric fatty diet
Dietary Supplement: ultra-high-caloric carbohydrate-rich diet — see arm/group description
  Arms: ultra-high-caloric carbohydrate-rich diet

SUMMARY:
The LIPCAL-ALS study (NCT02306590) has provided preliminary evidence that a high-caloric nutrition might prolong survival in fast-progressing ALS patients. Since increasing the amount of calories of the intervention might possibly increase the beneficial effect, the investigators seek to investigate whether an ultra-high caloric diet (UHCD), featuring the double amount of calories compared to LIPCAL-ALS, will be well tolerated by ALS patients and may serve as an intervention for a potential LIPCALII study. For this purpose, the investigators will compare two different UHCDs (one fat-rich and one carbohydrate-rich) with regard to safety and tolerability over a time frame of 4 weeks. A third group will receive the original diet from LIPCAL, and a fourth group will receive no intervention (control group).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Amyotrophic Lateral Sclerosis (ALS) according to the revised version of the El Escorial criteria (Ludolph et al. 2015)
* Slope of ALS Functional Rating Scale Revised (ALSFRS-R) of >0.25 points per month at baseline visit based on the formula (48 - score at baseline visit) / (time between date of first symptom and baseline visit)
* stable on standard therapy riluzole (100 mg/day) for at least 4 weeks
* capable of thoroughly understanding all information given and giving full informed consent according to good clinical practice (GCP)

Exclusion Criteria:

* already taking any dietary supplements
* participation in another clinical trial within the preceding 8 weeks
* tracheostomy or assisted ventilation of any type which exceeds 23 hours per day
* pregnancy or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events and Serious Adverse Events | 4 weeks
  Incidence of Adverse Events and Serious Adverse Events
Laboratory values | 4 weeks
  Incidence of abnormalities in clinical laboratory assessments, vital signs and physical examinations

SECONDARY OUTCOMES:
Appetite | 2 weeks; 4 weeks
  Change of Appetite-Score (Council of Nutrition appetite questionnaire, CNAQ) compared to baseline; values 8-40; higher values mean better appetite
Eating Habits | 2 weeks; 4 weeks
  Change in eating habits as evaluated by a standardized questionnaire (Ulmer eating habits questionnaire); descriptive information and evaluation; no overall score
Taste of Intervention | 2 weeks; 4 weeks
  taste of intervention (visual analogous scale); values 1-9, higher values mean better taste
Body Weight | 2 weeks; 4 weeks
  change of body weight compared to baseline
Biomarkers | 4 weeks
  change of neurofilament light chains (NfL) in serum
Adverse Events and Serious Adverse Events | 6 weeks
  Incidence of Adverse Events and Serious Adverse Events (evaluation via phone call 2 weeks after intervention was finished)
ALSFRS-R | 4 weeks
  change of Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) compared to baseline; values 0-48; higher values mean less impairment

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Dorst, PD Dr., Principal Investigator — University of Ulm
Locations (1):
- University of Ulm, Department of Neurology, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be available beginning 3 months and ending 5 years following article publication. Data will be shard with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims in the approved proposal. Proposals should be directed to johannes.dorst@uni-ulm.de; to gain access, data requestors will need to sign a data acess agreement. The study protocol will be available for 5 years at htpps://www.uniklinik-ulm.de/neurologie.html.
Supporting Information: Study Protocol
Time Frame: 3 month after publication until 5 years after publication
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims in the approved proposal. Proposals should be directed to johannes.dorst@uni-ulm.de; to gain access, data requestors will need to sign a data acess agreement.
URL: https://www.uniklinik-ulm.de/neurologie.html

REFERENCES:
- [Background] Ludolph A, Drory V, Hardiman O, Nakano I, Ravits J, Robberecht W, Shefner J; WFN Research Group On ALS/MND. A revision of the El Escorial criteria - 2015. Amyotroph Lateral Scler Frontotemporal Degener. 2015;16(5-6):291-2. doi: 10.3109/21678421.2015.1049183. Epub 2015 Jun 29. No abstract available. PMID 26121170